CLINICAL TRIAL: NCT06198842
Title: Clinical Open-label Phase 2 Study of Low Dose Treosulfan Based Conditioning Regimen Efficacy in Hematopoietic Stem Cell Transplantation With Post-transplant Cyclophosphamide for Children Nijmegen Breakage Syndrome
Brief Title: Low Dose Treosulfan Based Conditioning Regimen and PTCy in HSCT for Nijmegen Breakage Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Treo-NBS 2023
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Nijmegen Breakage Syndrome
MeSH Terms: conditions — Nijmegen Breakage Syndrome | interventions — treosulfan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental): Fludarabine 150mg/m2 (days -6, -5, -4, -3, -2) Treosulfan 21g/m2 (days -6, -5, -4) Thymoglobulin (Genzyme) 5mg/kg (days -5, -4) Rituximab 100mg/m2 (day -1) Cyclophosphamide 50mg/kg (days +3, +4)
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — Treosulfan 21mg/m2 (days -6, -5, -4)

SUMMARY:
The aim of the current study is to evaluate the safety and efficacy of low dose treosulfan based conditioning regimen in HSCT with post-transplant cyclophosphamide in Nijmegen breakage syndrome

DETAILED DESCRIPTION:
Nijmegen breakage syndrome (NBS) is a DNA repair disorder. The only curative option for combine immunodeficiency in NBS is allogeneic hematopoietic stem cell transplantation (HSCT). Standard myeloablative conditioning regimens in DNA repair disorders lead to increased morbidity and mortality after HSCT. Low doses of alkylators are used to reduce toxicity rates, which, however, increase the risks of mixed chimerism and graft failure. The data of treosulfan usage in NBS are sparse. To evaluate the safety and efficacy of low dose treosulfan based conditioning regimen in NBS, treosulfan 21g/m2 in combination with fludarabine 150mg/mg, thymoglobulin (Genzyme) 5mg/kg and rituximab 100mg/m2 will be used from day -6 to -1 day, followed by stem cell infusion and post-transplant cyclophosphamide 25mg/kg/day (+3,+4 day) for GVHD prophylaxis. The primary endpoint is event-free survival, where graft failure, death, and malignancies are considered as events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 3 months and < 21 years
2. Patients diagnosed with NBS eligible for an allogeneic HSCT
3. Signed written informed consent signed by a parent or legal guardian

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years after HSCT
  Events: graft failure, death, malignancies

SECONDARY OUTCOMES:
Overall survival | 3 years after HSCT
Cumulative incidence of engraftment | 100 days
Cumulative incidence of graft failure | 3 years
Cumulative incidence of viral infections | 1 year
Cumulative incidence of acute graft versus host disease | 1 year
Cumulative incidence of chronic graft versus host disease | 3 years
Incidence of early organ toxicity | 100 days
Cumulative incidence of transplant related mortality | 3 years
Incidence of long-term toxicity | 3 years
  malignancies, non-malignant complications

CONTACTS AND LOCATIONS:
Locations (1):
- HSCT department, Moscow, Russia